CLINICAL TRIAL: NCT00463541
Title: An Open-label Study of the Efficacy and Safety of 5 and 10mg VESIcare® (Solifenacin Succinate) in Patients With Overactive Bladder Symptoms VOLT: VESIcare® Open-Label Trial
Brief Title: Open-label Study of the Efficacy and Safety of VESIcare® in Patients With Overactive Bladder Symptoms
Acronym: VOLT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 905-UC-007
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Urinary Bladder, Overactive
Keywords: Urinary Bladder, Overactive; Urgency; VESIcare®; Solifenacin succinate
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: solifenacin succinate

INTERVENTIONS:
Drug: solifenacin succinate — oral
  Other Names: VESIcare (R); YM905

SUMMARY:
To evaluate the safety and efficacy of solifenacin succinate in subjects with overactive bladder symptoms (urgency, with or without urge incontinence, usually with frequency and nocturia).

DETAILED DESCRIPTION:
Study included a 24 week extension that did not occur due to FDA approval of the product.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of OAB (urgency, with or without urge incontinence, usually with frequency and nocturia) for ≥3 or more months.
* Patients may be included if they are on another OAB medication; however, patients must washout from other OAB medications for at least 7 days prior to receiving solifenacin succinate. Previous non-drug treatment of OAB is allowed if it has been established at least 4 weeks prior to study entry and is continued throughout the study.

Exclusion Criteria:

* -Significant stress incontinence or mixed stress/urge incontinence where stress is the predominant factor
* Evidence of urinary tract infection; chronic inflammation such as interstitial cystitis and bladder stones
* Clinically significant outflow obstruction (benign prostatic hyperplasia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2225 (Actual)
Dates: Start 2004-06; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of 5 and 10mg solifenacin succinate in patients with OAB symptoms | Weeks 4, 8 and 12

SECONDARY OUTCOMES:
Percentage of patients satisfied with 5mg treatment | Week 12
Percentage of patients obtaining additional benefit with increase to 10mg dose | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (174):
- United States (174):
  - Bay Minette, Alabama
  - Birmingham, Alabama
  - Decatur, Alabama
  - Huntsville, Alabama
  - Oro Valley, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Buena Park, California
  - Corte Madera, California
  - Culver City, California
  - Fresno, California
  - Fullerton, California
  - Huntington Beach, California
  - Long Beach, California
  - Los Angeles, California
  - Mission Viejo, California
  - Modesto, California
  - Oceanside, California
  - Orange, California
  - Paramount, California
  - Pomona, California
  - Sacramento, California
  - San Bernadino, California
  - San Diego, California
  - Torrance, California
  - Tustin, California
  - Upland, California
  - Vista, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Fort Collins, Colorado
  - Wheat Ridge, Colorado
  - Avon, Connecticut
  - Hartford, Connecticut
  - Wilmington, Delaware
  - Brandon, Florida
  - Coral Gables, Florida
  - Coral Springs, Florida
  - Delray Beach, Florida
  - Fort Myers, Florida
  - Ft.Lauderdale, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Merritt Island, Florida
  - Miami, Florida
  - Okeechobee, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Royal Palm Beach, Florida
  - Tampa, Florida
  - Wellington, Florida
  - Albany, Georgia
  - Atlanta, Georgia
  - Conyers, Georgia
  - Decatur, Georgia
  - Marietta, Georgia
  - Roswell, Georgia
  - Snellville, Georgia
  - Woodstock, Georgia
  - Chicago, Illinois
  - Evanston, Illinois
  - Greenville, Illinois
  - Libertyville, Illinois
  - Mattoon, Illinois
  - Park Ridge, Illinois
  - Indianapolis, Indiana
  - Mason City, Iowa
  - Arkansas City, Kansas
  - Newton, Kansas
  - Shawnee, Kansas
  - Topeka, Kansas
  - Wichita, Kansas
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Glen Burnie, Maryland
  - Milford, Massachusetts
  - Watertown, Massachusetts
  - Battle Creek, Michigan
  - Dearborn, Michigan
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Kalamazoo, Michigan
  - Saint Clair Shores, Michigan
  - Saint Louis Park, Minnesota
  - Gulfport, Mississippi
  - Jackson, Mississippi
  - Independence, Missouri
  - Jackson, Missouri
  - Kansas City, Missouri
  - Liberty, Missouri
  - Manchester, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Missoula, Montana
  - Omaha, Nebraska
  - Henderson, Nevada
  - Reno, Nevada
  - East Orange, New Jersey
  - Englewood, New Jersey
  - Fair Lawn, New Jersey
  - New Brunswick, New Jersey
  - Perth Amboy, New Jersey
  - Princeton, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Brooklyn, New York
  - Lake Success, New York
  - Liverpool, New York
  - Mineola, New York
  - New York, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - The Bronx, New York
  - Asheboro, North Carolina
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Columbus, North Carolina
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - McConnelsville, Ohio
  - Mentor, Ohio
  - Painesville, Ohio
  - Zanesville, Ohio
  - Norman, Oklahoma
  - Tulsa, Oklahoma
  - Bend, Oregon
  - Portland, Oregon
  - Woodburn, Oregon
  - Allentown, Pennsylvania
  - Bala-Cynwyd, Pennsylvania
  - Beaver, Pennsylvania
  - Bensalem, Pennsylvania
  - Bethel Park, Pennsylvania
  - Camp Hill, Pennsylvania
  - Dauphin, Pennsylvania
  - Duncansville, Pennsylvania
  - Elkins Park, Pennsylvania
  - Harrisburg, Pennsylvania
  - Philadelphia, Pennsylvania
  - Phoenixville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Williamsport, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Bartlett, Tennessee
  - Greeneville, Tennessee
  - Johnson City, Tennessee
  - Murfreesboro, Tennessee
  - Nashville, Tennessee
  - New Tazewell, Tennessee
  - Austin, Texas
  - Corsicana, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Salt Lake City, Utah
  - Sandy City, Utah
  - Charlottesville, Virginia
  - Hampton, Virginia
  - Vienna, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Huntington, West Virginia

REFERENCES:
- [Background] Capo' JP Jr, Laramee C, Lucente V, Fakhoury A, Forero-Schwanhaeuser S. Solifenacin treatment for overactive bladder in Hispanic patients: patient-reported symptom bother and quality of life outcomes from the VESIcare Open-Label Trial. Int J Clin Pract. 2008 Jan;62(1):39-46. doi: 10.1111/j.1742-1241.2007.01644.x. Epub 2007 Nov 23. PMID 18036164
- [Background] Mallett V, Burks D, Garely AD, Smith N. Solifenacin treatment for overactive bladder in black patients: patient-reported symptom bother and health-related quality of life outcomes. Curr Med Res Opin. 2007 Apr;23(4):821-31. doi: 10.1185/030079907x178847. PMID 17407639
- [Background] Garely AD, Kaufman JM, Sand PK, Smith N, Andoh M. Symptom bother and health-related quality of life outcomes following solifenacin treatment for overactive bladder: the VESIcare Open-Label Trial (VOLT). Clin Ther. 2006 Nov;28(11):1935-46. doi: 10.1016/j.clinthera.2006.11.010. PMID 17213014
- [Background] Garely AD, Lucente V, Vapnek J, Smith N. Solifenacin for overactive bladder with incontinence: symptom bother and health-related quality of life outcomes. Ann Pharmacother. 2007 Mar;41(3):391-8. doi: 10.1345/aph.1H581. Epub 2007 Mar 6. PMID 17341526
- [Background] Sand PK, Steers WD, Dmochowski R, Andoh M, Forero-Schwanhaeuser S. Patient-reported most bothersome symptoms in OAB: post hoc analysis of data from a large, open-label trial of solifenacin. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jun;20(6):667-75. doi: 10.1007/s00192-009-0840-y. Epub 2009 Mar 10. PMID 19434385
- [Derived] Capo' JP, Lucente V, Forero-Schwanhaeuser S, He W. Efficacy and tolerability of solifenacin in patients aged >/= 65 years with overactive bladder: post-hoc analysis of 2 open-label studies. Postgrad Med. 2011 Jan;123(1):94-104. doi: 10.3810/pgm.2011.01.2250. PMID 21293089